CLINICAL TRIAL: NCT00806169
Title: Intravitreal Combination Therapy Using Triamcinolone and Bevacizumab Improves Vision in Patients With Diabetic Retinopathy
Brief Title: Combined Triple Therapy in Diabetic Retinopathy (DRP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Michael Koss, PI, Johann Wolfgang Goethe University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-KTDRP-2008
Record Dates: First submitted 2008-12-04; First posted 2008-12-10 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Macular Edema; Diabetic Retinopathy
Keywords: combined therapy; DRP; efficacy; safety; sustainability; macular edema due to DRP
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy | interventions — Triamcinolone; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): group I (n=17) nonproliferative DR and ischemic maculopathy
  Interventions: Drug: triamcinolone and bevacizumab
- 2 (Experimental): group II (n=38) nonproliferative DR without ischemic maculopathy
  Interventions: Drug: triamcinolone and bevacizumab
- 3 (Experimental): group III (n=18) proliferative DR with or without ischemic maculopathy
  Interventions: Drug: triamcinolone and bevacizumab

INTERVENTIONS:
Drug: triamcinolone and bevacizumab

SUMMARY:
The aim of this pilot study was to investigate the effects of an intravitreal combination therapy using triamcinolone and bevacizumab in patients with macular edema due to diabetic retinopathy.

DETAILED DESCRIPTION:
This prospective, monocenter pilot case series was conducted between May 2006 and November 2008. Patients were included because of DME and signs of pre- and early proliferation because of diabetic retinopathy.73 eyes of 56 patients were included, all of which had signed an informed consent to perform a pharmacosurgical procedure consisting of a 23 gauge core Pars Plana Vitrectomy (sutureless single stitch sclerotomy, cutter with 300 cuts/minute) with removement of 1.5ml vitreous and substitution with 1ml BSS, 8mg triamcinolone, and 1.25 mg bevacizumab. At baseline and follow-up, the best corrected visual acuity (BCVA; 6 m Snellen), and intraocular pressure (IOP; Goldmann tonometry), and central macular thickness (optical coherence tomography) were determined. In addition, the need for further treatment and adverse events were monitored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetic retinopathy

  * macular edema more than 200 micron
  * vitreous bleeding because of angiography documented NVEs NVDs, based on the definitions of ETDRS

Exclusion Criteria:

* Prior intraocular injection within 4 months
* Core or complete vitrectomy
* History of glaucoma or ocular hypertension
* Presence of iris neovascularization
* Significant media opacity
* Monocularity and pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | Day of exam

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Vitreoretinal Surgery, Frankfurt am Main, Hesse, Germany